CLINICAL TRIAL: NCT00002915
Title: A PHASE I AND PHARMACOLOGICAL STUDY OF PENCLOMEDINE (NSC#338720, IND#43409) ADMINISTERED DAILY BY MOUTH FOR FIVE CONSECUTIVE DAYS IN PATIENTS WITH ADVANCED SOLID TUMOR MALIGNANCIES
Brief Title: Penclomedine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065290; P30CA006973 (NIH); JHOC-9637; NCI-T96-0031
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — penclomedine

INTERVENTIONS:
Drug: penclomedine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of penclomedine in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of oral penclomedine that can be administered daily for 5 days every 4 weeks in patients with advanced solid tumor malignancies. II. Describe and quantitate the toxic effects of penclomedine administered on this schedule in these patients. III. Study the clinical pharmacology and metabolism of penclomedine on this schedule, and seek pharmacodynamic correlates of pharmacologic parameters with clinical endpoints. IV. Study the bioavailability of oral penclomedine, and qualitatively compare metabolite profiles produced following oral and intravenous administration in these patients. V. Seek preliminary evidence of therapeutic activity of penclomedine in patients with advanced cancer.

OUTLINE: This is a dose-escalation study to estimate the maximum tolerated dose (MTD) of penclomedine. Cohorts of 3-6 patients are treated at escalating doses until the MTD is reached. Patients receive oral penclomedine for 5 consecutive days every 4 weeks. If tumor progression or unacceptable toxicity is documented during any treatment course, the patient is removed from study. A total of 10 patients will be treated at the dose determined to be the MTD (the recommended phase II dose).

PROJECTED ACCRUAL: An estimated 20 patients will be accrued over approximately 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically documented solid tumor that is refractory to conventional therapy or for which no conventional treatment exists No primary or secondary brain tumor No CNS disease or treatment-related CNS dysfunction No bone metastases involving 4 or more sites

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: At least 8 weeks Hematopoietic: Absolute neutrophil count greater than 1,500 Platelet count greater than 100,000 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Other: No active infection No history of egg protein allergy No prior gastric or small intestine resection or clinical evidence of malabsorption No history of medical, neurologic, or psychiatric disorder No concomitant medical problem unrelated to the malignancy that precludes study compliance or increases treatment risk No pregnant women Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No more than 4 courses of combination chemotherapy that included an alkylating agent, cisplatin, or carboplatin (applies once grade 1 or worse myelosuppression is reported on this study) No prior mitomycin or nitrosoureas At least 28 days since chemotherapy No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to wide ports involving pelvis or 20% of bone marrow At least 28 days since large-field radiotherapy No concurrent radiotherapy Surgery: At least 14 days since major surgery Other: No bone marrow transplantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-12

CONTACTS AND LOCATIONS:
Overall Officials: Ross C. Donehower, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States